CLINICAL TRIAL: NCT03686345
Title: Prospective Evaluation of a Continuation Therapy With Midostaurin in Adult Patients With Core-binding Factor Leukemia and Integrated Genetic Analysis: a Multi-center Phase II Study
Brief Title: Midostaurin Associated With Standard Chemotherapy in Patients With Core-binding Factor Leukemia
Acronym: AML FLT3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: didn't reach the primary endpoint
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REL-AML 001/2017; 2017-002094-18 (EudraCT Number)
Record Dates: First submitted 2018-07-04; First posted 2018-09-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Core Binding Factor Acute Myeloid Leukemia (CBF-AML)
Keywords: Midostaurin; Chemotherapy; Relapse Incidence; Overall Survival; Disease Free Survival; Minimal Residual Disease monitoring
MeSH Terms: interventions — midostaurin

STUDY DESIGN:
Intervention Model Description: Core binding factor acute myeloid leukemia (CBF-AML) patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Core binding factor acute myeloid leukemia (CBF-AML) (Experimental): Patients must have an unequivocal diagnosis of de novo-CBFL, prior to start midostaurin, documented by rearrangement of Core Binding Factor (CBF) genes, namely AML1-ETO and CBFB-MYH11. The experimental arm involves the administration of Midostaurin orally 50 mg (two 25 mg tablets) twice a day, from the end of induction chemotherapy, for 14 days. Patients should take Midostaurin at approximately 12 hours intervals. During all consolidation cycles, Midostaurin 50 mg (two 25 mg tablets) is administered orally twice a day, on days 8-21. Patients in complete remission after 3 cycles of remission consolidation therapy, will receive Midostaurin continuation therapy for 12 months. Midostaurin 50 mg (two 25 mg tablets) will be given orally twice a day for 12 months.
  Interventions: Drug: Midostaurin

INTERVENTIONS:
Drug: Midostaurin — Midostaurin associated with standard chemotherapy in patients with core-binding factor leukemia

SUMMARY:
The purpose of this single-arm, open label, phase-II trial, is to determine whether the association of Midostaurin to standard induction, consolidation therapy and in maintenance therapy as single agent, is effective in decrease relapse incidence, in patients with CBF-AML. The single-arm, open label, phase-II study is based on data obtained from previous clinical and pre-clinical studies, obtained by use of Midostaurin in patients with Acute Myeloid Leukemia (with or without FLT3 mutations) and in patients with Mast cell disorders (characterized by mutations in the C-KIT gene). The investigators believe that Midostaurin, associated with standard therapy Anthracycline/AraC Induction, to the consolidation regimen with high doses of araC and maintenance therapy to single agent in patients with acute myeloid leukemia core-binding factor can significantly reduce the incidence of recurrence of the disease, occurring in 40-50% of cases treated with standard therapy

DETAILED DESCRIPTION:
In this prospective, Interventional, Single-Arm, Open-Label, Phase-II Trial aims at demonstrating a decrease in the 2-year Relapse Incidence (RI) and in the 2-year Cumulative Relapse Incidence among the Midostaurin-treated patients compared to a cohort of historical controls. The investigators established that a 20% net reduction in the 2-year RI may be a clinically significant goal. So the investigators set our RI objective at 28%. Furthermore, the investigators will assess if the experimental treatment may obtain an increased 5-years Overall, Disease-Free and Event free Survival. The safety profile of Midostaurin given in combination with induction and consolidation chemotherapy and as a single agent in maintenance in CBFL patients will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures.
* Patients must be 18 to 65 years of age at the time of signing informed consent.
* Patients must have an unequivocal diagnosis of de novo-CBFL, prior to start midostaurin, documented by rearrangement of Core Binding Factor (CBF) genes, namely AML1-ETO and CBFB-MYH11, either with observation of t(8;21)(q22;q22) or inv(16)(p13; q32)/t(16;16)(p13; q32) by conventional cytogenetics or hybridization techniques or detection of fusion genes by PCR-polymerase chain reaction
* Patients must be fit to receive an anthracycline/AraC-based induction therapy (i.e. Ara-C 100 mg/m2 or 200 mg/m2 i.v. day, by continuous infusion for 7 days and Idarubicin 12 mg/m2 i.v. day or daunomycin 60 mg/m2 on days 1, 3 and 5)
* Patients must have an ECOG-Eastern Cooperative Oncology Group Performance Status of ≤ 2.
* Patients must have Total Bilirubin ≤ 1.5 x ULN, and AST or ALT ≤ 2.5 x ULN.
* Patients must have Serum Creatinine ≤ 1.5 x ULN.
* Women of child-bearing potential must have a negative pregnancy test before starting the protocol.

Exclusion Criteria:

* Prior therapy for AML with the following exceptions:

  1. emergency leukapheresis
  2. emergency treatment for hyperleukocytosis with hydroxyurea for ≤ 7 days
* Central nervous system involvement
* Presence of any uncontrolled bacterial, viral or fungal infection
* Known human immunodeficiency virus (HIV) positive
* An active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection. Patients whose disease is controlled under antiviral therapy should not be excluded.
* Presence of other active malignancies
* QTc > 470 msec (Bazett formula) on screening ECG
* Presence of significant uncontrolled or active cardiovascular disease, specifically including, but not restricted to:

  1. Myocardial infarction, unstable angina and/or congestive heart failure within 3 months prior to randomization
  2. History of clinically significant (as determined by the treating physician) atrial arrhythmia or any ventricular arrhythmia
  3. Uncontrolled hypertension
  4. Taking medications that are known to be associated with Torsades de Pointes.
* History of hypersensitivity to any drugs or metabolites of similar chemical classes as the study treatment.
* Pregnancy statements and contraception requirements:

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 4 months after stopping medication. Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject
* Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system, or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should also add a barrier method of contraception, particularly as it is currently unknown whether midostaurin may reduce the effectiveness of hormonal contraceptives. Sexually-active males unless they use a condom during intercourse with females of reproductive potential or pregnant women and for at least 4 months after stopping treatment to avoid conception or embryo-fetal harm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Relapse Incidence | 2 years
  To show that the percentage of relapsed patients is 28% or below

SECONDARY OUTCOMES:
Overall survival | 5 years
  To determine overall survival from achievement of first complete remission
Safety assessment - Frequency and severity of adverse events | Up to 30 days after last dose of study drug
  Incidence of toxicity, defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03. Frequency and severity of adverse events will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. An adverse event is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after patient's signed informed consent has been obtained.
Disease-free survival | 5 years
  To determine disease-free survival from achievement of first complete remission
Event-free survival | 5 years
  To determine event-free survival from diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Cà Granda - Niguarda S.C: Ematologia, Milan, Italy

REFERENCES:
- [Background] Cairoli R, Gatti A, Grillo G, Stefanucci MR, Di Camillo B, Fumagalli M, Krampera M, Nadali G, Zappasodi P, Borlenghi E, Todisco E, Ubezio M, Bernardi M, Molteni A, Basilico C, Turrini M, Greco R, Mancini V, Riva M, Bernasconi DP, Brando B, Veronese SM, Beghini A. Efficacy of Midostaurin Combined With Intensive Chemotherapy in Core Binding Factor Leukemia: A Phase II Clinical Trial. Am J Hematol. 2025 Feb;100(2):346-349. doi: 10.1002/ajh.27547. Epub 2024 Dec 10. PMID 39659145